CLINICAL TRIAL: NCT06034587
Title: A Prospective, Longitudinal, Intraindividual Clinical Study in Keloid With Multimodal Ultrasound Assessment
Brief Title: Multimodal Ultrasound Imaging Assessment on Keloid
Status: Completed | Type: Observational
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Wang Zhigang, chief physician, Chongqing Medical University
Other Study IDs: CQMUSAZL0619
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Keloid
Keywords: multimodal ultrasound; shear wave elastography; microvessel imaging
MeSH Terms: conditions — Keloid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- good response group of treated keloids: The Vancouver Scar Scale (VSS) is the most established questionnaire used for the evaluation of pathological scarring. This scale evaluates aspects of scar vascularity, pigmentation, pliability, and height, with the scoring system ranging from 0 to 15, where 0 is the least severe and 15 is the most severe.All the keloids in the study were classified into three categories based on the VSS score: mild (0-5), moderate (6-9), and severe (10-15).
  For treatment assessment, investigators further divided the treated participants into two groups: a good response group (showing an improvement of 5 or more points in the VSS score) and a poor response group (less than 5 points improvement in the VSS score)
  Interventions: Diagnostic Test: multimodal ultrasound; Radiation: radioisotope applicator therapy
- poor response group of treated keloids: The Vancouver Scar Scale (VSS) is the most established questionnaire used for the evaluation of pathological scarring. This scale evaluates aspects of scar vascularity, pigmentation, pliability, and height, with the scoring system ranging from 0 to 15, where 0 is the least severe and 15 is the most severe. All the keloids in the study keloids were classified into three categories based on the VSS score: mild (0-5), moderate (6-9), and severe(10-15).
  For treatment assessment, investigators further divided the treated participants into two groups: a good response group (showing an improvement of 5 or more points in the VSS score) and a poor response group (less than 5 points improvement in the VSS score)
  Interventions: Diagnostic Test: multimodal ultrasound; Radiation: radioisotope applicator therapy

INTERVENTIONS:
Diagnostic Test: multimodal ultrasound — An Aixplorer ultrasound machine (SuperSonic Imaging, Ltd, Aixen-Provence, France), equipped with AngioPLUS(AP) and shear wave elastography(SWE) functions, was used for all examinations using a 4-15MHz linear probe.AP function can detect microvessels of lesions,SWE can evaluate the stiffness of lesions and high frequency ultrasound can measure the thickness and volume of keloid.
Radiation: radioisotope applicator therapy — The radioisotope applicator therapy utilized 90Sr-90Y(0094SR814975) isotope, customized by the China Atomic Energy Research Institute. The element therapy instrument used had overall dimensions of 2.8cm x 2.8cm, with an effective treatment area of 2.0cm x 2.0cm. It delivered a radiation dose of 5.0Gy/h. Each patient received superficial radiation therapy through a single 90Sr source, administered in repeated doses. The isotope therapy instrument was customized to fit the exact size of the keloid, ensuring coverage the irradiation range extending 0.5cm beyond the keloid's edge. During treatment, the surface of the applicator was aligned with the irradiated area and directly contact the surface of the keloid tissue. The treatment was carried out low-dose irradiation method, over 5 sessions, with each session delivering a dose of 2Gy. Each irradiation lasted for 25min.

SUMMARY:
Skin keloids are common dermatological conditions that can lead to physical limitations, functional impairments, and deformities. Beyond the physiological implications, the aesthetic ramifications of keloids can also result in significant psychological distress, including anxiety and depression, causing both physical and emotional suffering to the affected individuals. The incidence of keloids is high, characterized by their chronicity, resistance to treatment, and high recurrence rate. They have become one of the most challenging conditions to treat across burn surgery, plastic surgery, and dermatology disciplines. The lack of standardized clinical treatment guidelines globally, combined with an absence of a well-defined standardized evaluation system, means that the effectiveness of various treatments is not consistently and objectively assessed, creating significant challenges in clinical applications. This project integrates traditional high-frequency ultrasound with cutting-edge technologies like real-time shear wave elastography and ultra-micro blood flow imaging. By using multimodal ultrasound, investigators aim to observe the therapeutic response of 90Sr-90Y patch treatment on skin keloids. Investigators seek to determine the objectivity and quantification role of multimodal ultrasound data and indicators in assessing keloid severity, including blood flow information and elasticity hardness. Another goal is to obtain quantitative data on keloid thickness, volume, stiffness, and microvascular distribution before and after treatment to monitor the therapy response. This would address the current limitations of subjective keloid scoring scales. It would also serve as an objective assessment standard for precise diagnosis, treatment, and follow-up of keloids in a clinical setting, thereby standardizing the clinical diagnosis and treatment of keloids.

DETAILED DESCRIPTION:
Currently, no one-size-fits-all approach exists and a universally accepted, standardized evaluation and treatment protocol remains elusive, making it challenging to determine which method is the most effective. Commonly used methods for assessing keloids, such as the Vancouver Scar Scale (VSS) and the Patient and Observer Scar Assessment Scale (POSAS), rely heavily on subjective evaluations based on observer perception and patient-reported experiences. These methods lack objective quantitative evaluation indicators and the ability to visualize subcutaneous tissues, limiting their individual clinical applicability. The Vancouver Scar Scale (VSS) is the most established questionnaire used for the evaluation of pathological scarring. This scale evaluates aspects of scar vascularity, pigmentation, pliability, and height, with the scoring system ranging from 0 to 15, where 0 is the least severe and 15 is the most severe. In the study, keloids were classified into three categories based on the VSS score: mild (0-5), moderate (6-9), and severe (10-15).

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 16 years and above
* Outpatients with no received any treatment in previous 6 months
* Willing to participate in this trial and have signed an informed consent form

Exclusion Criteria:

* Pregnant or breastfeeding women
* patients with malignant tumors, hypertension, diabetes, skin rupture, skin infection which may influence keloid healing and other dermatologic diseases

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 34 outpatients (mean age 43 ± 10.4 years, 14 male, 20 female) with untreated 63 keloids in different anatomical locations and 63 corresponding normal skin sites was performed
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Change in stiffness measured by SWE | from baseline to 6 months
  The difference of stiffness in good response group and poor response group
Change in microvessel signal grade measured by AP | from baseline to 6 months
  The difference of microvessel signal grade in good response group and poor response group
Change in thickness measured by high frequency ultrasound | from baseline to 6 months
  The difference of thickness in good response group and poor response group

CONTACTS AND LOCATIONS:
Overall Officials: Wang Zhigang, Study Chair — Chongqing Medical University
Locations (1):
- The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dirrichs T, Quack V, Gatz M, Tingart M, Rath B, Betsch M, Kuhl CK, Schrading S. Shear Wave Elastography (SWE) for Monitoring of Treatment of Tendinopathies: A Double-blinded, Longitudinal Clinical Study. Acad Radiol. 2018 Mar;25(3):265-272. doi: 10.1016/j.acra.2017.09.011. Epub 2017 Nov 16. PMID 29153963
- [Result] DeJong H, Abbott S, Zelesco M, Spilsbury K, Ziman M, Kennedy BF, Martin L, Wood FM. Objective quantification of burn scar stiffness using shear-wave elastography: Initial evidence of validity. Burns. 2020 Dec;46(8):1787-1798. doi: 10.1016/j.burns.2020.05.009. Epub 2020 May 19. PMID 32534890
- [Result] Schwaiger H, Reinholz M, Poetschke J, Ruzicka T, Gauglitz G. Evaluating the Therapeutic Success of Keloids Treated With Cryotherapy and Intralesional Corticosteroids Using Noninvasive Objective Measures. Dermatol Surg. 2018 May;44(5):635-644. doi: 10.1097/DSS.0000000000001427. PMID 29701618
- [Result] Nast A, Gauglitz G, Lorenz K, Metelmann HR, Paasch U, Strnad V, Weidmann M, Werner RN, Bauerschmitz J. S2k guidelines for the therapy of pathological scars (hypertrophic scars and keloids) - Update 2020. J Dtsch Dermatol Ges. 2021 Feb;19(2):312-327. doi: 10.1111/ddg.14279. Epub 2020 Oct 4. No abstract available. PMID 33015930
- [Result] Yang Y, Wang L, Yan F, Xiang X, Tang Y, Zhang L, Liu J, Qiu L. Determination of Normal Skin Elasticity by Using Real-time Shear Wave Elastography. J Ultrasound Med. 2018 Nov;37(11):2507-2516. doi: 10.1002/jum.14608. Epub 2018 Mar 25. PMID 29575120
- [Result] Yang Y, Qiu L, Wang L, Xiang X, Tang Y, Li H, Yan F. Quantitative Assessment of Skin Stiffness Using Ultrasound Shear Wave Elastography in Systemic Sclerosis. Ultrasound Med Biol. 2019 Apr;45(4):902-912. doi: 10.1016/j.ultrasmedbio.2018.11.015. Epub 2019 Jan 18. PMID 30665723
- [Result] Tsai WY, Hsueh YY, Chen PY, Hung KS, Huang CC. High-Frequency Ultrasound Elastography for Assessing Elastic Properties of Skin and Scars. IEEE Trans Ultrason Ferroelectr Freq Control. 2022 Jun;69(6):1871-1880. doi: 10.1109/TUFFC.2022.3154235. Epub 2022 May 26. PMID 35201987
- [Result] Guo R, Xiang X, Wang L, Zhu B, Cheng S, Qiu L. Quantitative Assessment of Keloids Using Ultrasound Shear Wave Elastography. Ultrasound Med Biol. 2020 May;46(5):1169-1178. doi: 10.1016/j.ultrasmedbio.2020.01.010. Epub 2020 Feb 13. PMID 32063394
- [Result] Reinholz M, Schwaiger H, Poetschke J, Epple A, Ruzicka T, Von Braunmuhl T, Gauglitz GG. Objective and subjective treatment evaluation of scars using optical coherence tomography, sonography, photography, and standardised questionnaires. Eur J Dermatol. 2016 Dec 1;26(6):599-608. doi: 10.1684/ejd.2016.2873. PMID 27762215
- [Result] Elrefaie AM, Salem RM, Faheem MH. High-resolution ultrasound for keloids and hypertrophic scar assessment. Lasers Med Sci. 2020 Mar;35(2):379-385. doi: 10.1007/s10103-019-02830-4. Epub 2019 Jun 25. PMID 31240510
- [Result] DeJong H, Abbott S, Zelesco M, Spilsbury K, Martin L, Sanderson R, Ziman M, Kennedy BF, Wood FM. A Novel, Reliable Protocol to Objectively Assess Scar Stiffness Using Shear Wave Elastography. Ultrasound Med Biol. 2020 Jul;46(7):1614-1629. doi: 10.1016/j.ultrasmedbio.2020.03.003. Epub 2020 May 5. PMID 32386847
- [Result] Xu C, Ting W, Teng Y, Long X, Wang X. Laser Speckle Contrast Imaging for the Objective Assessment of Blood Perfusion in Keloids Treated With Dual-Wavelength Laser Therapy. Dermatol Surg. 2021 Apr 1;47(4):e117-e121. doi: 10.1097/DSS.0000000000002836. PMID 33795568
- [Result] Son Y, Phillips EON, Price KM, Rosenberg LZ, Stefanovic B, Wolfe CM, Shaath TS, Om A, Cohen GF, Gunjan A. Treatment of keloids with a single dose of low-energy superficial X-ray radiation to prevent recurrence after surgical excision: An in vitro and in vivo study. J Am Acad Dermatol. 2020 Nov;83(5):1304-1314. doi: 10.1016/j.jaad.2020.06.023. Epub 2020 Jun 12. PMID 32540415
- [Result] Tang Y, Cheng S, Tang X, Guo R, Zhang L, Qiu L. Quantification of skin lesions using high-frequency ultrasound and shear wave elastography in port-wine stain patients: a clinical study. Ann Transl Med. 2019 Dec;7(24):803. doi: 10.21037/atm.2019.12.57. PMID 32042819
- [Result] Xiang X, Yan F, Yang Y, Tang Y, Wang L, Zeng J, Qiu L. Quantitative Assessment of Healthy Skin Elasticity: Reliability and Feasibility of Shear Wave Elastography. Ultrasound Med Biol. 2017 Feb;43(2):445-452. doi: 10.1016/j.ultrasmedbio.2016.10.002. Epub 2016 Dec 2. PMID 27919522
- [Result] Poetschke J, Schwaiger H, Gauglitz GG. Current and Emerging Options for Documenting Scars and Evaluating Therapeutic Progress. Dermatol Surg. 2017 Jan;43 Suppl 1:S25-S36. doi: 10.1097/DSS.0000000000000698. PMID 27153039
- [Derived] Zhou L, Zhou Q, Zheng C, Wang Z, Rao M. Multimodal ultrasound assessment for monitoring keloid severity and treatment response. Sci Rep. 2025 Mar 12;15(1):8568. doi: 10.1038/s41598-025-91111-y. PMID 40074795